**NCT No: Not assigned** 

Document date: April 3, 2021

Validation of Therapeutic Effects of Cefaly on Insomnia by Neuroimaging and Polysomnography Analyses: a single site, single-armed exploratory study

## **Statistical Analysis Plan**

- 1) At baseline, the demographic data of the patients will be analyzed with descriptive statistics (age, gender, education years, height and weight)
- 2) Changes of Pittsburgh sleep index, Insomnia severity index, and Epworth sleepiness scale, Polysomnography measures, Neuroimaging parameters between baseline and after 4 weeks of intervention will be analyzed with Wilcoxon's signed rank test.